CLINICAL TRIAL: NCT00377078
Title: Use of Recombinant Human Lactoferrin in Long-Term Care Patients With Feeding Tubes to Manage Post-Antibiotic Colonization and Infection With Clostridium Difficile
Brief Title: Use of Recombinant Human Lactoferrin in Long-Term Care Patients With Feeding Tubes With Clostridium Difficile.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Johns Hopkins University (Other)
Collaborators: Ventria Bioscience (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: CP-VB-04-02
Record Dates: First submitted 2006-09-14; First posted 2006-09-15 (Estimated); Last update posted 2006-09-15 (Estimated); Status verified 2006-09

CONDITIONS: Clostridium Difficile
Keywords: recombinant human lactoferrin

INTERVENTIONS:
Drug: recombinant human lactoferrin

SUMMARY:
Primary objective of this pilot study is to evaluate the effect of recombinant human lactoferrin on the rate of infection with Clostridium difficile in long-term care patients supported by enteral feeding requiring broad spectrum antibiotics.

DETAILED DESCRIPTION:
This study is a prospective, randomized, double blind, placebo controlled comparison.

Product to be tested: Lactoferrin (human) derived from rice.

Amount, dosage, route of administration, duration:Subjects will receive 3 grams of lactoferrin every 24 hours in the flush solution for the automated enteric feeding system. Dosing will begin with antibiotic dosing and continue for 8 weeks following the initial dose of antibiotic. If there is a change/adjustment in the antibiotics or initiation of another course of antibiotic therapy during the study period, blood and stool samples will be taken as an additional study point, but there will be no extension of the 8 weeks of study material administration.

Objectives: To test the use of lactoferrin (human) derived from rice in the management of post-antibiotic colonization with Clostridium difficile and the resulting inflammation reaction in the intestine in long-term care patients on enteral feeding.

Clinical Endpoints:

C. difficile antigen status change Diarrhea (2 or more loose stools, conforming to container, in 24 hours)

Clinical Markers:

C. difficile toxin status change Stool and serum proinflammatory and anti-inflammatory cytokines

1 antitrypsin serum and stool cRP - serum WBC - blood

Study Groups:

All patients on enteral feeding by gastrostomy, naso-gastric, or jejunostomy tubes.

At first antibiotic treatment (after start of study), subjects will be randomized to study treatment

Test: Recombinant human lactoferrin from rice in 50 mM NaCl in enteral feeding flush. 5 mg/mL lactoferrin in 600 mL 0.3% (50 mM) saline administered every 24 hours of the 8 weeks of the study period.

Controls: 600 mL 0.3% (50 mM) saline

All material for test and control flushing fluid will be supplied by Ventria Bioscience in containers labeled with the patient study number, enteral feeding system flush, expiration date and sponsor name. Codes will be held by Ventria and not broken until 30 patients are completed. A sealed copy of the code will be available to the principal investigator. In case of adverse events the code can be broken at the request of the principal investigator.

Preparation:

One bottle of flush solution powder is dissolved in 600 mL of water. The 600 mL of flush is used in a 24 hour period as the automatic flush by the standard enteral feeding pumps used. If there is flush material remaining at the end of a cycle, it will be administered as a bolus dose if less than 200 mL.

Subjects: Thirty patients will be enrolled with intent to treat in a masked, randomized, placebo controlled study. All subjects will be in the long-term care facility at Johns Hopkins Bayview Medical Center.

Inclusion Criteria

* Patients in long-term care facility, Ventilator Rehabilitation Unit (VRU) (Plaza) at the John Burton Care Center of the Johns Hopkins Bayview Medical Center.
* Nutrition via gastrostomy, naso-gastric or jejunostomy enteral feeding system.
* Patients with supplemental oral intake, but primary nutrition via gastrostomy/jejunostomy tube.
* Patients with colostomies are also allowed
* Not currently on antibiotic therapy and no antibiotics within 10 days.
* Patient is negative for Clostridium difficile antigen in screen
* Patient, guardian or health care agent willing to give informed consent.

Exclusion Criteria

* Patients who will only receive vancomycin, linezolid, or metronidazole as the antibiotic treatment, not broad spectrum antibiotics. All other antibiotics will qualify.
* Patients with illeostomies.
* Patients who have signs or symptoms of C. difficile infection; such as diarrhea (two or more liquid stools in a 24-hour period) and elevated WBC (more than 15,000/mm3).
* Known allergy to rice or rice products.

Additionally, the principal investigator may declare any patient ineligible if severity of illness may limit adequate time for follow-up data collection.

Study Procedures:All patients (new or current if they have been antibiotic treatment free for 10 days) negative for C. difficile on the VRU at the John Burton Care Center on enteral feeding will be invited to participate in the study. New patients are screened for C. difficile as part of admitting procedures; current patients will be screened for current C. difficile antigen status. Patients or guardian of patients interested in participation will be asked to sign an informed consent. When patient requires the first treatment with a broad spectrum antibiotic, they will be randomized into the study.

Study material will be administered via the flush cycle of the enteral feeding system. The typical daily flush is 600 mL of diluted saline. The study material will be in one third normal saline, approximately 0.3% or 50 mM with or without lactoferrin.

The recombinant human lactoferrin from rice will be at 5 mg/mL.

Study material will be used in the flush cycle, 600 mL per day, beginning on the first day of antibiotic treatment until 8 weeks following the final dose of antibiotic.

At entry into the study, patients will have blood and stool samples taken to assay for:

C. difficile antigen and toxin C. difficile bacterial culture, an aliquot of stool and all recovered organisms will be frozen for future analysis.

Serum and stool cytokines cRP - c reactive protein - blood

1 antitrypsin stool and blood White blood cell count and differential

Patients who have a positive C. difficile antigen at time zero will be exited from the study and will not be considered in the intent to treat analysis.

Samples will be taken again to assay for the above markers at two and six weeks after the start of antibiotic treatment, and at 8 weeks post antibiotics initiation or at exit from the study period. A stool sample will be collected weekly, in addition to the regular study time points. This sample will be frozen for future analysis.

Patients will be monitored daily during the study for occurrence of diarrhea throughout the study period. The definition of diarrhea will be that a stool flows to the shape of the container.

If a second course of antibiotics is required during the 8 week post antibiotic period, samples will be taken for assay of the study markers at that time and the study course will continue, but not be extended.

Patients who become positive for C. difficile will remain in the study until they require treatment for C. difficile. At initiation of treatment for C. difficile, study samples will be collected and the patient will be exited from the study, but included in the analysis. Patients who are C. difficile antigen positive will remain in the study until a positive test for C. difficile toxin A or B is confirmed.

Statistical Analyses: Data will be summarized as the number and percent of patients that convert from a negative to a positive C. difficile antigen and the number and percent of patients with reported diarrhea at any time. The number of days that subjects are diarrhea-free out of the 8-week study period will also be recorded. These data will be analyzed by a comparison of rates using Fisher's Exact Test with 95% confidence intervals.

Due to the small number of subjects in the study, the goal will be to identify trends rather than statistical significance

ELIGIBILITY:
Inclusion Criteria:

* Patients in long-term care facility, Ventilator Rehabilitation Unit (VRU) (Plaza) at the John Burton Care Center of the Johns Hopkins Bayview Medical Center.
* Nutrition via gastrostomy, naso-gastric or jejunostomy enteral feeding system.
* Patients with supplemental oral intake, but primary nutrition via gastrostomy/jejunostomy tube.
* Patients with colostomies are also allowed
* Not currently on antibiotic therapy and no antibiotics within 10 days.
* Patient is negative for Clostridium difficile antigen in screen
* Patient, guardian or health care agent willing to give informed consent.

Exclusion Criteria:

* Patients who will only receive vancomycin, linezolid, or metronidazole as the antibiotic treatment, not broad spectrum antibiotics. All other antibiotics will qualify.
* Patients with illeostomies.
* Patients who have signs or symptoms of C. difficile infection; such as diarrhea (two or more liquid stools in a 24-hour period) and elevated WBC (more than 15,000/mm3).
* Known allergy to rice or rice products.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2005-10; Study Completion 2007-10

PRIMARY OUTCOMES:
Subjects receive 3 grams of lactoferrin in a flush solution for the automated enteric feeding system.
Dosing will begin with antibiotic dosing

CONTACTS AND LOCATIONS:
Overall Officials: William B Greenough, III, MD, Principal Investigator — Johns Hopkins University; Delia Bethell, Ph.D., Study Director — Ventria Bioscience; Delia Bethell, Ph.D., Study Chair — Ventria Bioscience
Locations (1):
- Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States